CLINICAL TRIAL: NCT02419430
Title: Mindfulness Based Resilience Training for Employees at Mayo Clinic
Brief Title: Mindfulness Based Resilience Training
Acronym: MBRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Cynthia M. Stonnington, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-001492
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Stress, Psychological
Keywords: well-being; stress; resilience; self-compassion
MeSH Terms: conditions — Stress, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MBRT ClassRoom and Phone Application (Active Comparator): MBRT ClassRoom and Phone Application
  Interventions: Behavioral: MBRT ClassRoom and Phone Application
- Phone application only (Active Comparator): Phone application only
  Interventions: Behavioral: Phone application only
- Questionnaires (Active Comparator): Questionnaires
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: MBRT ClassRoom and Phone Application — 2 hours/week for 6 week, in classroom intervention involving mindfulness based resilience training.focused on mindfulness and self-compassion training, including body awareness, breath awareness, mindful movement, awareness of thoughts, and awareness of emotion. Core concepts included: normalizing experience of stress and changing one's relationship with an experience; learning to be a compassionate observer of self in order to appreciate the moment; recognizing undue efforts to control something that has already happened; shifting attention to felt body sense and away from the narrative; and redirecting attention to a value as a way of evoking positive states that enhance the present moment experience. Participants also use the smartphone to track their sleep and subjective well-being.
  Arms: MBRT ClassRoom and Phone Application
Behavioral: Phone application only — Participants will track their sleep and subjective well-being and also choose one of the following weekly challenges, which is completed via smartphone interactions:
  * Joys of Life
  * Count your blessings
  * Think differenc, feel better
  * Exercising --> Happier
    + Exercising --> Sleep
  * Pre-Sleep routine
  * Eat that frog
  * Mindful Meditation
  Arms: Phone application only
Behavioral: Questionnaires — At baseline, immediately after the last MBRT session (6 weeks) and again at 3 and 6 months, all participants will complete questionnaires, including: 1) WHO-5 Well-Being Index; 2) DASS-21; 3) VAS-Fatigue; 4) MBI-Human Services version; 5) Self-Compassion Scale; 6) Connor-Davidson 2-item resilience scale; 7) Compassion to others scale.
  Arms: Questionnaires

SUMMARY:
The investigators aim to evaluate the Mindfulness Based Resilience Training (MBRT) intervention for Mayo Clinic employees in order to provide evidence for improved ability to cope with stress and decreased work-related burnout and stress-related symptoms as a result of MBRT training. In addition, the investigators aim to compare the effects of MBRT + smartphone sleep feedback, a smartphone resilience intervention + smartphone sleep feedback, or waitlist control +smartphone sleep feedback in a randomized clinical trial in a sample of 75 Mayo Clinic employees.

DETAILED DESCRIPTION:
The investigators aim to compare the effects of MBRT + smartphone sleep feedback, a smartphone resilience intervention + smartphone sleep feedback, or waitlist control +smartphone sleep feedback in a randomized clinical trial in a sample of 75 Mayo Clinic employees. Specific self-report outcomes include: well-being, stress, anxiety, depression, fatigue, resilience, self-compassion, and burn-out, assessed at pre-, post- and 3-month followup. Objective outcomes, derived from smartphone-driven self-monitoring, include sleep quality and emotional experiencing, assessed throughout the six-week intervention period. The investigators will explore whether changes in objectively measured sleep quality and emotional experiencing will mediate treatment effects on self-report outcomes. The investigators will also explore whether treatment effects are more robust in self-selected versus randomized groups by drawing on the investigators' existing data.

ELIGIBILITY:
Inclusion:

1. Stress subscale of the DASS-21 needs to be a score 5 or greater and
2. Must have a smart Phone, and
3. Ability to attend at least 5 complete sessions.

Exclusion :

1. Stress subscale of the DASS-21 less than 5.
2. Must have a smart Phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in scores using the DASS-21(Depression Anxiety and Stress Scales) questionnaire | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stonnington, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States